CLINICAL TRIAL: NCT04283578
Title: Oxytocin Treatment in Neonates and Infants Aged From 0 to 3 Months With Prader-Willi Syndrome : a Study of Safety and Efficacy on Oral and Social Skills and Feeding Behavior of Intranasal Administration of Oxytocin vs Placebo
Brief Title: Oxytocin Treatment in Neonates and Infants With Prader-Willi Syndrome
Acronym: OTBB3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: International Clinical Trials Association (Other); Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/15/7825
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): intranasal administration of OT
  Interventions: Drug: OT; Drug: Placebo comparator
- Placebo (Placebo Comparator): intranasal administration of placebo
  Interventions: Drug: OT; Drug: Placebo comparator

INTERVENTIONS:
Drug: OT — One group will receive OT for 4 weeks, then placebo or OT for 8 weeks
  Other Names: oxytocin
Drug: Placebo comparator — One group will receive Placebo for 4 weeks, then Placebo or OT for 8 weeks.

SUMMARY:
Prospective, randomized, placebo-controlled, double-blind part of the phase III trial to assess the safety and efficacy of 4 weeks oxytocin (OT) administration on oral and social skills in neonates/infants with Prader-Willi Syndrome (PWS) aged less than 3 months at inclusion. Phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female neonate or infant, with PWS genetically confirmed.
2. Age <92 days (plus a tolerance of up to 8 days maximum) (for preterm infants, born before 37 weeks amenorrhea, corrected age will be applied).
3. Signed informed consent obtained from the parents/holders of parental authority.
4. Parents willing and able to comply with all study procedures.

Exclusion Criteria:

* 1. Neonate or infant currently admitted to the emergency care unit for ongoing life-threatening comorbidities like severe respiratory, cardiovascular or neurological abnormalities.

  2. Neonate or infant with prolongation of the QT interval. 3. Neonate or infant without medical insurance. 4. Neonate or infant with hypersensitivity to oxytocin or excipients of the product.

  5. Neonate or infant with concomitant treatment prolonging QT interval 6. Neonate or infant with family history of genetic pathology causing QT interval prolongation.

  7. Neonate or infant with hypokalemia (clinically relevant at the discretion of the doctor).

  8. Neonate or infant participating simultaneously in another interventional study.

  9. Neonates or infants whose parents' situations may jeopardize the interpretation of the results.

  10. Neonates or infants whose parents' refuse video recording, required to respond to the primary objective of the study.

Ages: 1 Day to 92 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Neonatal Oral-Motor Assessment Scale (NOMAS) scale | 4 weeks
  the score goes from 8 to 28, the higher the score meaning a worse outcome

SECONDARY OUTCOMES:
Ghrelin dosage | Day 0, Week 1 and week 4
  Concentration of ghrelin (unacylated/UAG and acylated/AG)
Oxytocin dosage | Day 0, week 4
  Plasma Oxytocin concentration
Proficiency score | Day 0, Week and week 4
  The volume of milk taken in the first five minutes of feeding

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- Cliniques Saint Luc, Brussels, Belgium
- France (5):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la Timone Enfant, Marseille
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Centre de réfrence Prader-Willi, Hospital of infants, Toulouse
- Klinik für Kinderheilkunde II, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borie AM, Dromard Y, Guillon G, Olma A, Manning M, Muscatelli F, Desarmenien MG, Jeanneteau F. Correction of vasopressin deficit in the lateral septum ameliorates social deficits of mouse autism model. J Clin Invest. 2021 Jan 19;131(2):e144450. doi: 10.1172/JCI144450. PMID 33232306